CLINICAL TRIAL: NCT07196683
Title: Regenerative Potentials of Mature Mandibular First Molars With Symptomatic Irreversible Pulpitis Enhanced With Different Scaffolds: A Randomized Controlled Trial
Brief Title: Regenerative Potentials of Mature Mandibular Molars With Symptomatic Irreversible Pulpitis Enhanced With Different Scaffolds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Abdel Hakim, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: New ENDO 5-5-1
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP)
Keywords: pulpotomy, regenerative pulpotomy, ascorbic acid-augmented PRF, tannic acid crosslinked-PRF

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ascorbic acid augmented PRF scaffold (Experimental)
  Interventions: Procedure: Regenerative pulpotomy
- Tannic acid cross linked PRF scaffold (Experimental)
  Interventions: Procedure: Regenerative pulpotomy
- PRF scaffold (Active Comparator)
  Interventions: Procedure: Regenerative pulpotomy

INTERVENTIONS:
Procedure: Regenerative pulpotomy — Regenerative pulpotomy combines the use of hydraulic calcium silicate based cements; MTA, together with biodegradable scaffolds such as PRF.
  Other Names: Vital pulp therapy; PRF pulpotomy

SUMMARY:
The current study aims to assess the influence of different scaffolds on postoperative pain and success rate of pulpotomy in mandibular mature molars with symptomatic irreversible pulpitis

DETAILED DESCRIPTION:
The study aims to assess different scaffolds used in regenerative pulpotomy of mature permanent mandibular first molars diagnosed with symptomatic irreversible pulpitis and their influence on postoperative pain and clinical and radiographic success rate of pulpotomy. It also aims to correlate the level of inflammatory mediators in pulpal blood to the success rate of pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Age between 15-40 years.
* Males & Females.
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent (Appendix I).
* Mature mandibular fist molars:

  * Diagnosed clinically with symptomatic irreversible pulpitis and normal periapical tissue.
  * Giving a positive response to pulp sensitivity testing.
  * Having negative response to percussion.
  * Having normal radiographic appearance of periapical tissues.
  * Having bright red color of pulp tissue, with hemorrhage control within 10 mins, upon access cavity preparation.

Exclusion Criteria:

* Pregnant and lactating females.
* Patients with physical or mental handicapping conditions.
* Patients unwilling to participate in a 12-months follow up.
* Mandibular first molars with:

  * Immature roots.
  * Negative response to pulp sensitivity testing.
  * Positive response to percussion.
  * Radiographic evidence of periapical lesions, external or internal root resorption, vertical root fracture, or calcification.
  * Intraoral swelling or fistula.
  * Lack of pulpal bleeding, or inability to achieve hemostasis of the bleeding pulp within 10 mins, upon access cavity preparation.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 6, 12, 24, and 72 hours postoperatively
  measured using numerical rating scale

SECONDARY OUTCOMES:
Overall success rate | 1, 3, 6, 9 and 12 months postoperatively.
  Based on clinical and radiographic signs and symptoms
IL-8 and TNF-α levels in pulpal blood | Upon access cavity preparation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided